CLINICAL TRIAL: NCT06648096
Title: Phase Ib/II Study to Investigate the Safety and Efficacy of Afatinib When Administered As Therapy in Fanconi Anemia Patients with Unresectable and / or Metastatic Locoregionally Advanced Squamous Cell Carcinoma of the Oral Cavity, Oropharynx or Hypopharynx or Larynx.
Brief Title: Afatinib in Patients with Fanconi Anemia (FA) and Advanced Head and Neck Squamous Cell Carcinoma (HNSCC)
Acronym: AFAN
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: MFAR Clinical Research S.L. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRSSP-001; 2024-511477-29-00 (EU CTIS Number)
Record Dates: First submitted 2024-10-15; First posted 2024-10-18 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Fanconi Anemia; Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Fanconi Anemia; Squamous Cell Carcinoma of Head and Neck | interventions — Afatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Afatinib (Experimental): Afatinib starting at 20 mg (weeks 1-2), escalating to 30 mg after two weeks (weeks 3-4) and escalating to 40 mg after one month (week 5 - thereafter) if no hematologic or other relevant toxicities are observed (CTCAE V5.0 < grade 2)
  Interventions: Drug: Afatinib

INTERVENTIONS:
Drug: Afatinib — Afatinib starting at 20 mg (weeks 1-2), escalating to 30 mg after two weeks (weeks 3-4) and escalating to 40 mg after one month (week 5 - thereafter) if no hematologic or other relevant toxicities are observed (CTCAE V5.0 < grade 2)

SUMMARY:
This research study is a phase Ib/II, single-arm, non-randomized, non-blind, multicenter study designed to determine whether Afatinib is effective and safe in patients with locoregionally unresectable and / or metastatic HNSCC with Fanconi Anemia.

The main hypothesis, based on preclinical evidence, is that treatment with afatinib, an epithelial growth factor receptor (EGFR) tyrosine kinase inhibitor (TKI), could be an effective treatment option to control cancer for patients with FA - HNSCC.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent according to local guidelines, must be signed and dated by the participant and investigator prior to performing any protocol procedure.
2. Patient is ≥ 18 years of age.
3. Confirmed diagnosis of Fanconi anemia.
4. Histologically or cytologically confirmed unresectable or locoregionally advanced squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx, larynx, nasopharynx, paranasal sinuses or salivary glands. Patients with distal metastasis (M1, American Joint Cancer Committee (AJCC) 8th ed.) are also eligible.
5. Tumor not a candidate for resection prior to Afatinib due to technical inability to resect (tumor fixation / invasion in the skull base, cervical vertebrae, nasopharynx or fixed lymph nodes) and / or low surgical cure [T3-T4, N2-N3; , AJCC 8th ed.]).
6. Patients must have at least 1 measurable lesion by computed tomography (CT) scan or magnetic resonance imaging (MRI) as defined by RECIST v1.1.
7. Previous anticancer treatment is allowed if it ends 6 weeks or 5 half-lives, whichever is shorter, before the expected date of start of the study treatment.
8. Previous locoregional treatments such as radiotherapy are allowed.
9. Eastern Cooperative Oncology Group (ECOG) performance status < 2 at inclusion.
10. Adequate organ and bone marrow functions, as defined below:

    1. Neutrophils > 1000 cells / microliter.
    2. Platelets > 50,000 cells / microliter.
    3. Hemoglobin > 8 g / dL
    4. Creatinine < 1.5 x upper limit normal (ULN) with clearance > 50 mL / min.
    5. Total bilirubin < 1.5 x ULN. Note: patients with Gilbert's may be included with bilirubin <2 x ULN.
    6. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5 x ULN or < 5 ULN if liver metastases are present.
    7. International normalized ratio (INR) and prothrombin time (PT) <1.5 x ULN.
11. Female patients must either:

    1. Be of non-childbearing potential:

       Postmenopausal *(defined as at least 1 year without any menses) prior to screening , or Documented surgically sterile (e.g.hysterectomy, bilateral salpingectomy, bilateral oophorectomy, or bilateral tubal occlusion).

       *Those who are amenorrheic due to an alternative medical cause are not considered postmenopausal and must follow the criteria for childbearing potential subjects.

       OR
    2. If of childbearing potential:

    Agree not to try to become pregnant during the study and for at least 1 months after the final study drug administration, And have a negative urine or serum pregnancy test within 7 days prior to Day 1 (females with false positive results and documented verification of negative pregnancy status are eligible for participation), And if heterosexually active, agree to abstinence (if in line with the usual preferred lifestyle of the patient) or consistently use a condom plus 1 form of highly effective birth control per locally accepted standards starting at screening and throughout the study period and for at least 1 month after the final study drug administration.
12. Female patients must agree not to breastfeed or donate ovules starting at screening and throughout the study period, and for at least 1 month after the final study drug administration.
13. Male patients must not donate sperm starting at screening and throughout the study period, and for at least 1 month after the final study drug administration.
14. Male patients with a partner with childbearing potential, or who is pregnant or breastfeeding must agree to abstinence or use a condom plus 1 form of highly effective birth control throughout the study period and for at least 1 month after the final study drug administration.
15. Patient agrees not to participate in another interventional study while on treatment in the present study.

Exclusion Criteria:

1. Patients who are candidates for surgery with curative intent are not eligible.
2. Less than two weeks from surgical resection or other major surgical procedure at start of treatment. Planned surgery for other diseases.
3. Previous treatment with EGFR small molecule inhibitors, EGFR inhibitory antibodies and / or any investigational agents for the treatment of HNSCC within 4 weeks prior to the selection was not allowed.

   Note: Previous treatment with chemotherapy and/or radiotherapy is allowed.
4. Patient must have recovered from any previous treatment toxicity to Grade ≤ 2.
5. Existence of any other intercurrent malignant disease is not allowed within the previous 2 years to inclusion.

   Note: Patients with non melanoma skin cancer, curatively treated localized prostate cancer, or carcinoma in situ of any type (if complete resection was performed) are allowed.
6. Active severe Severe infectious disease in the 4 weeks prior to the initiation of study treatment, including . Known human immunodeficiency virus (HIV) infection or chronic Hepatitis B or C.
7. Patient has documented history of a cerebral vascular event (stroke or transient ischemic attack), or the following criteria for cardiac disease:

   1. Myocardial infarction or unstable angina pectoris within 6 months of enrollment.
   2. History of serious ventricular arrhythmia (ie, ventricular tachycardia or ventricular fibrillation), high-grade atrioventricular block, or other cardiac arrhythmias requiring antiarrhythmic medications (except for atrial fibrillation that is well controlled with antiarrhythmic medication); history of QT interval prolongation.
   3. New York Heart Association (NYHA) class III or greater congestive heart failure or left ventricular ejection fraction of < 40%.
8. Participants with QTc interval (corrected) > 470 msec at screening.
9. History of interstitial lung disease requiring corticosteroids or pneumonitis.
10. Gastrointestinal disorders that may interfere with the absorption of the study drug or chronic diarrhea.
11. Patient has known hypersensitivity to afatinib or to any excipient contained in the drug formulation.
12. Female patients who are or intend to be pregnant or breastfeeding during their participation in the study or 1 month after the final study drug administration.
13. Patients unable to comply with the protocol as determined by the investigator.
14. The patient is currently participating in another clinical trial that would interfere with the radiological imaging schedule or any other determinations required in this protocol.
15. Patient has other underlying medical conditions that, in the opinion of the investigator, would impair the ability of the patient to receive or tolerate the planned treatment and follow-up.
16. Patients with psychiatric disorders that may interfere with monitoring.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-11-08 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | At 9-months after the first dose of study treatment
  Assessed by the investigator through imaging follow-up (CT scan/MRI) using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. This will be considered as the percentage/proportion of patients with confirmed complete response (CR) or partial response (PR) as their overall best response throughout the first 9 months after the first dose of afatinib. Objective responses will be assessed locally by the investigator according to RECIST, V1.1, and indicating the change in size of tumors as compared with baseline, at the first dose of study treatment.

SECONDARY OUTCOMES:
Disease control rate (DCR) | Throughout the study period, at least 9 months
  Percentage/proportion of patients with complete response (CR) or partial response (PR), according to ORR definition for the trial, or maintained stable disease (SD) as their overall best response, assessed by imaging follow-up (CT scan/MRI) and RECIST V1.1 criteria. Stable disease should be maintained for at least 4 months to be considered as a DCR event.
Duration of response (DoR) | Throughout the study period, at least 9 months
  Time from first confirmed response (CR or PR), according to ORR definition for the trial, to the date of the documented progression of the disease (PD) as determined using RECIST V1.1 criteria or death due to any cause, whichever occurs first. Those patients with response and without PD or death event will be censored on the date of their last tumor assessment.
Disease-free survival (DFS) | Throughout the study period, at least 9 months
  Time from first dosing date to the date of PD /secondary primary tumor (SPT) according to RECIST V1.1. Patients alive and free of events at the date of the analysis will be censored at their last known tumor assessment. Patients who start a new treatment line without progression /SPT will be censored on the date of first dose of the subsequent anticancer treatment.
Overall survival (OS) | Throughout the study period, at least 9 months
  defined as the time elapsed from the first dose of study treatment until death from any cause. We will assess the median OS, estimated by Kaplan-Meier. Patients alive and free of events at the date of the analysis will be censored at their last known contact.
Patient reported health-related quality of life (HRQoL) QLQ-C30 | At baseline and every 8 weeks until tumor recurrence, approximately 9 months
  assessed through the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C30 (EORTC QLQ-C30), version 3. The endpoint will report a numerical value that ranges from 0 to 100. Higher values indicate better performances status for all items but for symptoms, in which higher indicates greater or stronger symptoms.
Patient reported health-related quality of life (HRQoL) QLQ-HN43 | At baseline and every 8 weeks until tumor recurrence, approximately 9 months
  assessed through the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire EORTC head and neck cancer specific complementary module QLQ-HN43. The endpoint will report a numerical value that ranges from 0 to 100. Higher values indicate better performances status for all items but for symptoms, in which higher indicates greater or stronger symptoms.
Patient reported health-related quality of life (HRQoL) EQ-5D | At baseline and every 8 weeks until tumor recurrence, approximately 9 months
  assessed through the EQ-5D Health Status Questionnaire. The endpoint will report a numerical value that ranges from 0 to 100. Higher values indicate better performances status for all items but for symptoms, in which higher indicates greater or stronger symptoms.
Rate of severe toxicities | Throughout the study period, at least 9 months
  Percentage of patients experiencing Grade 3-5 treatment-related Adverse events (AEs) ) assessed by national cancer institute (NCI) Common Terminology Criteria for Adverse Events CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Surrallés, M.D.; Ph.D., Study Chair — Sant Pau's Hospital Research Institute
Locations (2):
- Medizinische Hochschule Hannover, Hanover, Germany
- Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No
No individual patient data will be shared

REFERENCES:
- [Derived] Anguera G, Gallego O, Llobet M, Berga N, Moreno-Martinez ME, Leon X, Kratz C, Garcia-Escudero R, Minguillon J, Surralles J. Opening of a phase Ib/II study to investigate the safety and efficacy of Afatinib in patients with Fanconi anemia and unresectable locally advanced or metastatic head and neck squamous cell carcinoma. BMC Cancer. 2025 Aug 26;25(1):1374. doi: 10.1186/s12885-025-14619-6. PMID 40859225